CLINICAL TRIAL: NCT05052151
Title: Hemodynamic Effects of Low vs. High Dialysate Temperature or Bicarbonate Concentration in Chronic Hemodialysis Patients
Brief Title: Temperature and Bicarbonate: Hemodynamic Effects During Dialysis
Acronym: TURBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 23-06-21
Record Dates: First submitted 2021-08-26; First posted 2021-09-22 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2021-08

CONDITIONS: End Stage Renal Disease on Dialysis

STUDY DESIGN:
Intervention Model Description: The study will be a single-blinded, randomized, controlled, crossover study with each participant being his or her own control. Participants will be blinded to the intervention and the order of the interventions will be random.
  Participants will be randomized using bloc randomization. We will create two blocs with 8 participants in each. The four dialysis sessions will be conducted on the same weekday each week, which results in a 1-week wash-out period with standard dialysis treatment between interventions.
Who Masked: Participant
Masking Description: Temperature or bicarbonate settings will not be revealed to participants during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low temperature (Active Comparator): Dialysate temperature
  Interventions: Other: Low dialysate temperature
- High temperature (Active Comparator): Dialysate temperature
  Interventions: Other: High dialysate temperature
- Low bicarbonate (Active Comparator): Dialysate bicarbonate concentration
  Interventions: Other: Low dialysate bicarbonate concentration
- High bicarbonate (Active Comparator): Dialysate bicarbonate concentration
  Interventions: Other: High dialysate bicarbonate concentration

INTERVENTIONS:
Other: Low dialysate temperature — 35°C
  Arms: Low temperature
Other: High dialysate temperature — 37°C
  Arms: High temperature
Other: Low dialysate bicarbonate concentration — 30 mmol/L
  Arms: Low bicarbonate
Other: High dialysate bicarbonate concentration — 38 mmol/L
  Arms: High bicarbonate

SUMMARY:
To elucidate the role of dialysate temperature and bicarbonate on hemodynamic parameters, plasma pH and electrolytes that potentially mediate this effect, the investigators wish to conduct a single-blinded, randomized, controlled, crossover study, specifically examining the effects of

* A fixed low temperature dialysate of 35°C compared to a fixed dialysate temperature of 37°C.
* A low dialysate bicarbonate concentration of 30 mmol/L compared to a high dialysate bicarbonate concentration of 38 mmol/L.

DETAILED DESCRIPTION:
Background

Intradialytic hypotension (IDH) is a common complication of hemodialysis (HD) and is considered one of the most frequent complications with a prevalence between 10-12% depending on the definition of IDH (1). IDH has been associated with inefficient dialysis (2), vascular access thrombosis (3) and mortality (4,5).

Orthostatic hypotension (OH) is another common complication in HD with a prevalence around 42% in patients initiating HD treatment (6). OH is significantly associated with worse outcome in HD patients in terms of an increased two-year mortality (4) and increased risk of all-cause death (6).

Understanding the mechanisms underlying IDH and OH has the potential to optimize HD treatment, in order to minimize the occurrence of IDH and OH, potentially improving not only patient mortality and morbidity but also the everyday comfort of chronic HD patients when receiving dialysis treatment.

This study will investigate the hemodynamic effect of alterations in dialysate bicarbonate and dialysate temperature.

Dialysate temperature

Several clinical studies have examined the effect of low temperature dialysate (LTD) on IDH, but only few have examined the hemodynamic response in detail with intradialytic measurements of cardiac output (CO), central blood volume (CBV) and total peripheral resistance (TPR) (7-14). Generally, the studies confirm a blood pressure (BP) stabilizing effect of LTD, but diverse results are found on changes in CO, CBV and TPR. Some studies found greater increase in TPR during dialysis with LTD compared to a higher dialysate temperature (8,9,11,14). Other studies found that intradialytic CBV (7,12) and CO (12) improved considerably with LTD.

One previous study (14) examined OH in relation to use of LTD, but not with detailed intradialytic hemodynamic measurements. The study showed that both supine and upright mean arterial blood pressure (MAP) were significantly lower after dialysis with a dialysate temperature of 37°C compared to a dialysate temperature of 35°C. Furthermore, the increase in TPR was greater during dialysis with LTD.

Dialysate bicarbonate

Few studies have investigated the effect of dialysate bicarbonate (DB) concentration on intradialytic hemodynamics and results have been conflicting. Lower DB (from 32 to 26 mmol/L or a reduction of 6 mmol/L, respectively) was in two cross-over studies (15,16) shown to increase systolic BP (SBP) by approximately 5 mmHg, whereas a third study reported no significant effect on BP (17). One of these studies also found an increase in TPR with lower DB (16). IDH has been associated with lower DB in one of the previously mentioned cross-over studies (15), but this association was not found by Gabutti et al in 2005 (17) or in larger observational studies (17-19). Manipulation of DB inevitably affects plasma pH of the patient during dialysis. Thus, if pH decreases with DB-induced acidosis, hydrogen ions displace cations such as calcium from protein binding sites. DB-induced alkalosis on the other hand increases pH, which promotes increased protein binding, which decreases free cation levels. At the same time, intracellular sequestration of potassium at high pH levels has also been speculated to lower plasma potassium levels (20). Consequently, by changing DB a range of electrolytes including calcium are potentially affected which could impact neuromuscular function and thereby intradialytic hemodynamic parameters and the frequency of IDH and OH (17,21-26).

Hypotheses

Hemodialysis or hemodiafiltration (HdF) sessions with a decreased dialysate temperature (35°C vs. 37°C) or decreased DB concentration (30 mmol/L vs. 38 mmol/L) will have the following effects:

* An increase in SBP, MAP and orthostatic blood pressure (OBP).
* An increase in one or more of the following: Cardiac output (CO), total peripheral resistance (TPR), central blood volume (CBV), stroke volume (SV) and/or heart rate (HR).
* A decrease in the frequency of IDH and OH.

Study participants

Participants will be recruited from the maintenance HD and HdF population associated with the Department of Renal Medicine at Aarhus University Hospital in Denmark. These include the Dialysis Clinic at Aarhus University Hospital as the main hub and satellite dialysis clinics in Randers and Horsens.

Power and sample size

Measurements from 30 randomly selected HD patients in our clinic yielded SD = 23 mmHg for the difference between within-treatment changes in SBP (non-standardized conditions). Assuming a lower SD due to standardized BP-measurements and strict in- and exclusion criteria an SD = 12 mmHg was used as a reasonable estimate. Sample size calculation with Stata/IC 16.1 (StataCorp, 4905 Lakeway Dr, College Station, TX 77845, USA) using analysis for a one-sample mean test (t-test), assuming a minimal detectable difference in means (mean difference between the two within-treatment changes in SBP) = 10 mmHg; SD = 12 mmHg; two-sided significance level (alpha) = 0.05; power=0.80 resulted in 14 participants. However, to account for dropout of two participants, a sample size of 16 was chosen.

Dialysis machines, filters, and dialysate composition

Dialysis console Fresenius 5008F (Fresenius Medical Care, Bad Homburg, Germany) and HD or HdF filters regularly used for treatment of the patient will be used in all dialysis sessions.

The standard dialysate prescribed for each individual patient will be used in all dialysis sessions thereby maintaining similar composition regarding electrolytes such as sodium, potassium, calcium, magnesium and chloride. Bicarbonate concentration will only be adjusted in the sessions investigating low (30 mmol/L) and high (38 mmol/L) DB concentration, respectively. Dialysate will be prepared on-line by the dialysis machine. Blood flow rate and dialysate flow rate will be kept as usual and will remain equal in all sessions regardless of intervention. Ultrafiltration rate will be kept constant and equal in the two dialysis sessions. The same applies for the volume of substitution fluid in HdF.

Orthostatic hypotension (OH)

OH is defined as a reduction in SBP of at least 20 mmHg or in DBP of at least 10 mmHg within 3 minutes of standing (27).

Intradialytic hypotension (IDH)

IDH is defined as a decrease in SBP ≥20 mmHg or a decrease in MAP ≥10 mmHg associated with clinical events/symptoms (e.g. muscle cramps, abdominal discomfort, nausea or vomiting, dizziness or fainting, restlessness or anxiety, yawning or signing) and/or need for intradialytic interventions (Trendelenburg positioning, fluid administration, reduction in ultrafiltration rate, reduction of blood flow rate) or dialysis treatment cessation (28).

Intradialytic measurements

Cardiac output (CO) will be obtained by a previously validated ultrasound dilution technique using Hemodialysis Monitor HD03, Flow-QC tubing sets, and clip-on flow/dilution sensors from Transonic Systems Inc., Ithaca, NY, USA (29-32). The ultrasound sensors will be positioned on the arterial and venous Flow-QC tubing set using standard ultrasound gel to secure good contact. Access recirculation in the AV-fistula can invalidate CO-measurements. A built-in recirculation protocol will be used to check for access recirculation using injection of 10 mL isotonic saline into the venous blood line prior to the first CO-measurement. If recirculation is detected the dialysis needles will most likely be reinserted. CO will be measured in duplicate by injecting a bolus of 30 mL 37°C isotonic saline into the venous blood line within 5 seconds. If results deviate more than 15% a third measurement will be done. The mean of the two closest recordings will serve as the result. With the Transonic device intradialytic hemodynamic parameters are obtained at 10, 70, 130, 190, and 230 minutes. Patients will be lying in a supine position with the head elevated 20 degrees. Before each CO measurement HR and BP will be measured. MAP, TPR, and SV are derived by the following equations:

MAP = diastolic BP + 1/3 x (systolic BP - diastolic BP)

CO = SV x HR = MAP/TPR

CBV is defined as the volume of blood in the heart, lungs and great vessels and is estimated with the Transonic device based on the CO measurement.

Blood samples and handling of biological material

Following the same time pattern as the Transonic measurements an arterial blood gas will be drawn from the arterial cannula.

Eleven blood samples will be taken from the arterial blood line via the AV-cannula used for dialysis treatment. Four of the samples will be regular blood samples of 3-4 mL, whereas 7 of the samples will be arterial blood gases of 1 mL. Thus, per session 22 mL blood per participant is collected which adds up to a total of 88 mL for the entire study period. The purpose of this is to determine several essential parameters:

* Electrolytes such as calcium, magnesium, and potassium
* Acid-base status: pH, standard bicarbonate, standard base excess
* Hemoglobin, hematocrit
* Urea for the determination of Kt/V and URR.
* White cell count and C-reactive protein in the first blood sample in order to confirm the absence of infection

All blood samples will be transferred to the laboratory according to standard routine and analyzed according to current clinical standards at Department of Clinical Biochemistry, Aarhus University Hospital or local Department of Clinical Biochemistry normally servicing our satellite dialysis clinics in Randers and Horsens. Blood gas tests are analyzed using ABL blood gas analyzer (Radiometer, Radiometer Medical ApS, Brønshøj Denmark). All blood samples will be destroyed after analysis.

No samples will be stored in a biobank.

ELIGIBILITY:
Inclusion Criteria:

* Regular dialysis (HD or HDF) therapy for >3 months
* Age >18 years
* Stable and functional arteriovenous (AV)-fistula
* Able to achieve a dialysis blood flow > 250 mL
* Able to stand up for a minimum of 10 min
* Able to undergo a 4 hour dialysis session without eating, drinking or sleeping
* Proven cabable of cumulative ultrafiltration of 2% of end-dialytic weight (EDW)
* Able to give informed consent to participation in the study
* Hematocrit >30%
* BMI >18 and <35

Exclusion Criteria:

* Central venous catheter for HD or HDF
* Recirculation in AV-fistula
* Acute myocardial infarction within 3 months
* Atrial fibrillation
* Active malignant or infectious diseases
* Cerebrovascular incident within 3 months
* Pregnancy
* Alcohol or drug abuse
* History of interruptions during HD or untimely termination of HD treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Blood pressure (BP) | 4 weeks
  SBP (mmHg), Mean BP (mmHg) and Ortostatic BP (mmHg)

SECONDARY OUTCOMES:
Intradialytic cardiac output | 4 weeks
  CO (L/min)
Intradialytic total peripheral resistance | 4 weeks
  TPR (mmHg/(L/min))
Intradialytic stroke volume | 4 weeks
  SV (mL)
Intradialytic heart rate | 4 weeks
  HR (beats/min)
Intradialytic central blood volume | 4 weeks
  CBV (L)
Intradialytic mean arterial blood pressure | 4 weeks
  MAP (mmHg)
Plasma calcium | 4 weeks
  Calcium (mmol/L)
Plasma potassium | 4 weeks
  Potassium (mmol/L)
Plasma magnesium | 4 weeks
  Magnesium (mmol/L)
Intradialytic hypotension (IDH) | 4 weeks
  IDH frequency (number of events)
Ortostatic hypotension (OH) | 4 weeks
  OH frequency (number of events)

CONTACTS AND LOCATIONS:
Overall Officials: Niels H Buus, Professor, Study Chair — Department of Renal Medicine, Aarhus University Hospital; Jens D Jensen, MD, PhD, Study Chair — Department of Renal Medicine, Aarhus University Hospital; Ina H Jørgensen, Student, Principal Investigator — Department of Renal Medicine, Aarhus University Hospital; Jonas SK Jensen, Student, Principal Investigator — Department of Renal Medicine, Aarhus University Hospital; Christian D Peters, MD, PhD, Principal Investigator — Department of Renal Medicine, Aarhus University Hospital
Locations (1):
- Dialysis Clinic at Department of Renal Medicine, Aarhus University Hospital and affiliated dialysis clinics in Randers and Horsens, Aarhus, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuipers J, Verboom LM, Ipema KJR, Paans W, Krijnen WP, Gaillard CAJM, Westerhuis R, Franssen CFM. The Prevalence of Intradialytic Hypotension in Patients on Conventional Hemodialysis: A Systematic Review with Meta-Analysis. Am J Nephrol. 2019;49(6):497-506. doi: 10.1159/000500877. Epub 2019 May 24. PMID 31129661
- [Background] Ronco C, Brendolan A, Milan M, Rodeghiero MP, Zanella M, La Greca G. Impact of biofeedback-induced cardiovascular stability on hemodialysis tolerance and efficiency. Kidney Int. 2000 Aug;58(2):800-8. doi: 10.1046/j.1523-1755.2000.00229.x. PMID 10916105
- [Background] Chang TI, Paik J, Greene T, Desai M, Bech F, Cheung AK, Chertow GM. Intradialytic hypotension and vascular access thrombosis. J Am Soc Nephrol. 2011 Aug;22(8):1526-33. doi: 10.1681/ASN.2010101119. PMID 21803971
- [Background] Shoji T, Tsubakihara Y, Fujii M, Imai E. Hemodialysis-associated hypotension as an independent risk factor for two-year mortality in hemodialysis patients. Kidney Int. 2004 Sep;66(3):1212-20. doi: 10.1111/j.1523-1755.2004.00812.x. PMID 15327420
- [Background] Tisler A, Akocsi K, Borbas B, Fazakas L, Ferenczi S, Gorogh S, Kulcsar I, Nagy L, Samik J, Szegedi J, Toth E, Wagner G, Kiss I. The effect of frequent or occasional dialysis-associated hypotension on survival of patients on maintenance haemodialysis. Nephrol Dial Transplant. 2003 Dec;18(12):2601-5. doi: 10.1093/ndt/gfg450. PMID 14605284
- [Background] Sasaki O, Nakahama H, Nakamura S, Yoshihara F, Inenaga T, Yoshii M, Kohno S, Kawano Y. Orthostatic hypotension at the introductory phase of haemodialysis predicts all-cause mortality. Nephrol Dial Transplant. 2005 Feb;20(2):377-81. doi: 10.1093/ndt/gfh614. Epub 2004 Dec 23. PMID 15618243
- [Background] Beerenhout C, Dejagere T, van der Sande FM, Bekers O, Leunissen KM, Kooman JP. Haemodynamics and electrolyte balance: a comparison between on-line pre-dilution haemofiltration and haemodialysis. Nephrol Dial Transplant. 2004 Sep;19(9):2354-9. doi: 10.1093/ndt/gfh315. Epub 2004 Jul 20. PMID 15266029
- [Background] Yu AW, Ing TS, Zabaneh RI, Daugirdas JT. Effect of dialysate temperature on central hemodynamics and urea kinetics. Kidney Int. 1995 Jul;48(1):237-43. doi: 10.1038/ki.1995.289. PMID 7564084
- [Background] van der Sande FM, Wystrychowski G, Kooman JP, Rosales L, Raimann J, Kotanko P, Carter M, Chan CT, Leunissen KM, Levin NW. Control of core temperature and blood pressure stability during hemodialysis. Clin J Am Soc Nephrol. 2009 Jan;4(1):93-8. doi: 10.2215/CJN.01800408. Epub 2008 Oct 8. PMID 18842948
- [Background] Selby NM, Burton JO, Chesterton LJ, McIntyre CW. Dialysis-induced regional left ventricular dysfunction is ameliorated by cooling the dialysate. Clin J Am Soc Nephrol. 2006 Nov;1(6):1216-25. doi: 10.2215/CJN.02010606. Epub 2006 Oct 11. PMID 17699351
- [Background] Kaufman AM, Morris AT, Lavarias VA, Wang Y, Leung JF, Glabman MB, Yusuf SA, Levoci AL, Polaschegg HD, Levin NW. Effects of controlled blood cooling on hemodynamic stability and urea kinetics during high-efficiency hemodialysis. J Am Soc Nephrol. 1998 May;9(5):877-83. doi: 10.1681/ASN.V95877. PMID 9596086
- [Background] Hoeben H, Abu-Alfa AK, Mahnensmith R, Perazella MA. Hemodynamics in patients with intradialytic hypotension treated with cool dialysate or midodrine. Am J Kidney Dis. 2002 Jan;39(1):102-7. doi: 10.1053/ajkd.2002.29887. PMID 11774108
- [Background] Chesterton LJ, Selby NM, Burton JO, McIntyre CW. Cool dialysate reduces asymptomatic intradialytic hypotension and increases baroreflex variability. Hemodial Int. 2009 Apr;13(2):189-96. doi: 10.1111/j.1542-4758.2009.00355.x. PMID 19432693
- [Background] Jost CM, Agarwal R, Khair-el-Din T, Grayburn PA, Victor RG, Henrich WL. Effects of cooler temperature dialysate on hemodynamic stability in "problem" dialysis patients. Kidney Int. 1993 Sep;44(3):606-12. doi: 10.1038/ki.1993.287. PMID 8231034
- [Background] Gabutti L, Ferrari N, Giudici G, Mombelli G, Marone C. Unexpected haemodynamic instability associated with standard bicarbonate haemodialysis. Nephrol Dial Transplant. 2003 Nov;18(11):2369-76. doi: 10.1093/ndt/gfg383. PMID 14551368
- [Background] Gabutti L, Bianchi G, Soldini D, Marone C, Burnier M. Haemodynamic consequences of changing bicarbonate and calcium concentrations in haemodialysis fluids. Nephrol Dial Transplant. 2009 Mar;24(3):973-81. doi: 10.1093/ndt/gfn541. Epub 2008 Oct 8. PMID 18842671
- [Background] Gabutti L, Ross V, Duchini F, Mombelli G, Marone C. Does bicarbonate transfer have relevant hemodynamic consequences in standard hemodialysis? Blood Purif. 2005;23(5):365-72. doi: 10.1159/000087193. Epub 2005 Jul 27. PMID 16088104
- [Background] Tentori F, Karaboyas A, Robinson BM, Morgenstern H, Zhang J, Sen A, Ikizler TA, Rayner H, Fissell RB, Vanholder R, Tomo T, Port FK. Association of dialysate bicarbonate concentration with mortality in the Dialysis Outcomes and Practice Patterns Study (DOPPS). Am J Kidney Dis. 2013 Oct;62(4):738-46. doi: 10.1053/j.ajkd.2013.03.035. Epub 2013 May 24. PMID 23707043
- [Background] Viegas M, Candido C, Felgueiras J, Clemente J, Barros S, Farbota R, Vera F, Matos A, Sousa F. Dialysate bicarbonate variation in maintenance hemodiafiltration patients: Impact on serum bicarbonate, intradialytic hypotension and interdialytic weight gain. Hemodial Int. 2017 Jul;21(3):385-392. doi: 10.1111/hdi.12502. Epub 2016 Oct 20. PMID 27761981
- [Background] Heguilen RM, Sciurano C, Bellusci AD, Fried P, Mittelman G, Rosa Diez G, Bernasconi AR. The faster potassium-lowering effect of high dialysate bicarbonate concentrations in chronic haemodialysis patients. Nephrol Dial Transplant. 2005 Mar;20(3):591-7. doi: 10.1093/ndt/gfh661. Epub 2005 Feb 1. PMID 15687112
- [Background] Gabutti L, Salvade I, Lucchini B, Soldini D, Burnier M. Haemodynamic consequences of changing potassium concentrations in haemodialysis fluids. BMC Nephrol. 2011 Apr 6;12:14. doi: 10.1186/1471-2369-12-14. PMID 21470404
- [Background] Kyriazis J, Kalogeropoulou K, Bilirakis L, Smirnioudis N, Pikounis V, Stamatiadis D, Liolia E. Dialysate magnesium level and blood pressure. Kidney Int. 2004 Sep;66(3):1221-31. doi: 10.1111/j.1523-1755.2004.00875.x. PMID 15327421
- [Background] Elsharkawy MM, Youssef AM, Zayoon MY. Intradialytic changes of serum magnesium and their relation to hypotensive episodes in hemodialysis patients on different dialysates. Hemodial Int. 2006 Oct;10 Suppl 2:S16-23. doi: 10.1111/j.1542-4758.2006.00120.x. PMID 17022745
- [Background] Pakfetrat M, Roozbeh Shahroodi J, Malekmakan L, Zare N, Hashemi Nasab M, Hossein Nikoo M. Is there an association between intradialytic hypotension and serum magnesium changes? Hemodial Int. 2010 Oct;14(4):492-7. doi: 10.1111/j.1542-4758.2010.00477.x. PMID 20955283
- [Background] Kyriazis J, Glotsos J, Bilirakis L, Smirnioudis N, Tripolitou M, Georgiakodis F, Grimani I. Dialysate calcium profiling during hemodialysis: use and clinical implications. Kidney Int. 2002 Jan;61(1):276-87. doi: 10.1046/j.1523-1755.2002.00100.x. PMID 11786110
- [Background] Karamperis N, Sloth E, Jensen JD. The hemodynamic effect of calcium ion concentration in the infusate during predilution hemofiltration in chronic renal failure. Am J Kidney Dis. 2005 Sep;46(3):470-80. doi: 10.1053/j.ajkd.2005.05.022. PMID 16129209
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Kooman J, Basci A, Pizzarelli F, Canaud B, Haage P, Fouque D, Konner K, Martin-Malo A, Pedrini L, Tattersall J, Tordoir J, Vennegoor M, Wanner C, ter Wee P, Vanholder R. EBPG guideline on haemodynamic instability. Nephrol Dial Transplant. 2007 May;22 Suppl 2:ii22-44. doi: 10.1093/ndt/gfm019. No abstract available. PMID 17507425
- [Background] Krivitski NM, Depner TA. Cardiac output and central blood volume during hemodialysis: methodology. Adv Ren Replace Ther. 1999 Jul;6(3):225-32. doi: 10.1016/s1073-4449(99)70018-x. PMID 10452705
- [Background] Kisloukhine VV, Dean DA. Validation of a novel ultrasound dilution method to measure cardiac output during hemodialysis. ASAIO J. 1996 Sep-Oct;42(5):M906-7. doi: 10.1097/00002480-199609000-00125. PMID 8945018
- [Background] Tsutsui M, Matsuoka N, Ikeda T, Sanjo Y, Kazama T. Comparison of a new cardiac output ultrasound dilution method with thermodilution technique in adult patients under general anesthesia. J Cardiothorac Vasc Anesth. 2009 Dec;23(6):835-40. doi: 10.1053/j.jvca.2009.03.007. Epub 2009 May 22. PMID 19464193
- [Background] Moser M, Kenner T. Blood flow and blood volume determinations in aorta and in coronary circulation by density dilution. Basic Res Cardiol. 1988 Nov-Dec;83(6):577-89. doi: 10.1007/BF01906951. PMID 3223874
- [Background] Daugirdas JT. Second generation logarithmic estimates of single-pool variable volume Kt/V: an analysis of error. J Am Soc Nephrol. 1993 Nov;4(5):1205-13. doi: 10.1681/ASN.V451205. PMID 8305648
- [Background] Ayoub A, Finlayson M. Effect of cool temperature dialysate on the quality and patients' perception of haemodialysis. Nephrol Dial Transplant. 2004 Jan;19(1):190-4. doi: 10.1093/ndt/gfg512. PMID 14671056
- [Background] Sajadi M, Gholami Z, Hekmatpou D, Soltani P, Haghverdi F. Cold Dialysis Solution for Hemodialysis Patients With Fatigue: a Cross-over Study. Iran J Kidney Dis. 2016 Sep;10(5):319-324. PMID 27721231

DOCUMENTS (1):
  • Study Protocol (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT05052151/Prot_000.pdf